CLINICAL TRIAL: NCT05308810
Title: Evaluation of Postoperative Kidney Functions in Geriatric Patients Undergoing Major Gynecologic-Oncologic Surgery: A Retroceptive - Cohort Study
Brief Title: Postoperative Kidney Functions in Geriatric Major Gynecologic-Oncologic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Principal İnvestigator, Ankara City Hospital Bilkent
Other Study IDs: E1-22-2381
Record Dates: First submitted 2022-03-18; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Geriatrics; Acute Renal Injury; Gynecologic Surgery
Keywords: Geriatrics; Acute Renal Injury; Gynecologic Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Major Gynecologic- oncologic Surgery — Major Gynecologic-Oncologic surgery between january 2020 - january 2022

SUMMARY:
The increasing number of patients who develop perioperative acute kidney injury (AKI) is partly related to the aging population and the increasing number of individuals with chronic comorbidities, particularly those with premorbid chronic kidney disease. Anesthesiologists and surgeons will increasingly have to deal with such patients who are elderly and have comorbidities and require major surgery.

The aim of this study was to determine the incidence of postoperative acute kidney injury (primary aim) in patients aged 65 and over who underwent elective major gynecological-oncological surgery under general anesthesia in Ankara City Hospital Gynecology-Oncology Operating Room between January 2020-2022 and were followed up in the PACU in the postoperative period. To investigate risk factors and their results in a retrospective manner in line with the KDIGO criteria (secondary purpose).

ELIGIBILITY:
Inclusion Criteria:

* patients underwent major abdominal gynecologic oncologic surgery between January 2021 and January 2022
* followed in the PACU

Exclusion Criteria:

* Patients with inaccessible data and missing data

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — undergone major abdominal gynecologic oncologic surgery between
Study Population: patients underwent major abdominal gynecologic oncologic surgery and followed in the PACU between January 2021 and January 2022 at Ankara City hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
the incidence of the patients with AKI STAGE 1 | 48 hours after surgery
  AKI STAGE 1 : increase Cr ≥ 0.3 mg/dl or increase Cr to 1.5-1.9 times from baseline; or urine volume < 0.5 ml/kg/h for 6-12 hours
  AKI STAGE 2 :
  increase to 2-2.9 times from baseline; or urine volume < 0.5 ml/kg/h for ≥ 12 hours
  AKI STAGE 3 :
  increase Cr to ≥ 3 times from baseline; or increase Cr ≥ 4 mg/dl or initiation of renal replacement therapy or decrease in GFR to <35mL/min/1.73 m2 or urine volume < 0.3 ml/kg/h for ≥ 24 hours or Anuria for ≥ 12 hours
the incidence of the patients with AKI stage 2 | 48 hours after surgery
  AKI STAGE 1 : increase Cr ≥ 0.3 mg/dl or increase Cr to 1.5-1.9 times from baseline; or urine volume < 0.5 ml/kg/h for 6-12 hours
  AKI STAGE 2 :
  increase to 2-2.9 times from baseline; or urine volume < 0.5 ml/kg/h for ≥ 12 hours
  AKI STAGE 3 :
  increase Cr to ≥ 3 times from baseline; or increase Cr ≥ 4 mg/dl or initiation of renal replacement therapy or decrease in GFR to <35mL/min/1.73 m2 or urine volume < 0.3 ml/kg/h for ≥ 24 hours or Anuria for ≥ 12 hours
the incidence of the patients with AKI stage 3 | 48 hours after surgery
  AKI STAGE 1 : increase Cr ≥ 0.3 mg/dl or increase Cr to 1.5-1.9 times from baseline; or urine volume < 0.5 ml/kg/h for 6-12 hours
  AKI STAGE 2 :
  increase to 2-2.9 times from baseline; or urine volume < 0.5 ml/kg/h for ≥ 12 hours
  AKI STAGE 3 :
  increase Cr to ≥ 3 times from baseline; or increase Cr ≥ 4 mg/dl or initiation of renal replacement therapy or decrease in GFR to <35mL/min/1.73 m2 or urine volume < 0.3 ml/kg/h for ≥ 24 hours or Anuria for ≥ 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Postaci, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided